CLINICAL TRIAL: NCT03411525
Title: Provider, Patient, and Health System Effects of Provider Commitments to Choose Wisely
Brief Title: Effects of Provider Commitments to Choose Wisely
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Donaghue Medical Research Foundation (Other); Integrated Health Associates (Unknown)
Responsible Party: Principal Investigator, Jeffrey T. Kullgren, Assistant Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00112834
Record Dates: First submitted 2018-01-19; First posted 2018-01-26 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Health Services Misuse; Physician's Practice Patterns; Guideline Adherence; Unnecessary Procedures; Health Care Costs

STUDY DESIGN:
Intervention Model Description: Stepped wedge cluster randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Commitment invitation at time 1 (Experimental): In the stepped wedge cluster randomized design, the first clinic will remain in the control period (no intervention) for 1 month, followed by a 1 month transition period (where data will not be collected), before crossing over to the intervention period for 8 months.
  Interventions: Behavioral: Commitment Invitation for Clinicians (Clinician Intervention); Other: Health Education Materials to Patients (Patient Intervention)
- Commitment invitation at time 2 (Experimental): In the stepped wedge cluster randomized design, the second clinic will remain in the control period (no intervention) for 2 months, followed by a 1 month transition period (where data will not be collected), before crossing over to the intervention period for 7 months.
  Interventions: Behavioral: Commitment Invitation for Clinicians (Clinician Intervention); Other: Health Education Materials to Patients (Patient Intervention)
- Commitment invitation at time 3 (Experimental): In the stepped wedge cluster randomized design, the third clinic will remain in the control period (no intervention) for 3 months, followed by a 1 month transition period (where data will not be collected), before crossing over to the intervention period for 6 months.
  Interventions: Behavioral: Commitment Invitation for Clinicians (Clinician Intervention); Other: Health Education Materials to Patients (Patient Intervention)
- Commitment invitation at time 4 (Experimental): In the stepped wedge cluster randomized design, the fourth clinic will remain in the control period (no intervention) for 4 months, followed by a 1 month transition period (where data will not be collected), before crossing over to the intervention period for 5 months.
  Interventions: Behavioral: Commitment Invitation for Clinicians (Clinician Intervention); Other: Health Education Materials to Patients (Patient Intervention)
- Commitment invitation at time 5 (Experimental): In the stepped wedge cluster randomized design, the fifth clinic will remain in the control period (no intervention) for 5 months, followed by a 1 month transition period (where data will not be collected), before crossing over to the intervention period for 4 months.
  Interventions: Behavioral: Commitment Invitation for Clinicians (Clinician Intervention); Other: Health Education Materials to Patients (Patient Intervention)
- Commitment invitation at time 6 (Experimental): In the stepped wedge cluster randomized design, the sixth clinic will remain in the control period (no intervention) for 6 months, followed by a 1 month transition period (where data will not be collected), before crossing over to the intervention period for 3 months.
  Interventions: Behavioral: Commitment Invitation for Clinicians (Clinician Intervention); Other: Health Education Materials to Patients (Patient Intervention)
- Commitment invitation at time 7 (Experimental): In the stepped wedge cluster randomized design, the seventh clinic will remain in the control period (no intervention) for 7 months, followed by a 1 month transition period (where data will not be collected), before crossing over to the intervention period for 2 months.
  Interventions: Behavioral: Commitment Invitation for Clinicians (Clinician Intervention); Other: Health Education Materials to Patients (Patient Intervention)
- Commitment invitation at time 8 (Experimental): In the stepped wedge cluster randomized design, the eighth clinic will remain in the control period (no intervention) for 8 months, followed by a 1 month transition period (where data will not be collected), before crossing over to the intervention period for 1 month.
  Interventions: Behavioral: Commitment Invitation for Clinicians (Clinician Intervention); Other: Health Education Materials to Patients (Patient Intervention)

INTERVENTIONS:
Behavioral: Commitment Invitation for Clinicians (Clinician Intervention) — Clinicians will be invited to commit to follow 3 Choosing Wisely® recommendations. Those that choose to commit will sign a written document, appear on in-clinic posters along with their colleagues who have committed to the recommendations, have access to point-of-care Choosing Wisely® patient education handouts, and receive weekly emails with decision support resources.
Other: Health Education Materials to Patients (Patient Intervention) — During the intervention period, the letter and study information sheet that eligible patients will receive in advance of a scheduled appointment with a participating clinician will also be accompanied by a patient education handout from Consumer Reports that is publicly available and may be relevant to their health and health care. Specifically, patients with type 2 diabetes who are 65 and older will receive a handout about diabetes overtreatment, patients with insomnia or anxiety who are 65 and older will receive a handout about overuse of benzodiazepines and sedative-hypnotics, and male patients who are 75 and older with no history of prostate cancer will receive a handout about overuse of PSA tests to screen for prostate cancer.

SUMMARY:
Clinicians' decisions to order potentially unnecessary services -- such as those targeted in the Choosing Wisely® campaign -- are often affected by their high-pressure practice environments, which can make it hard to consistently avoid ordering low-value care. The field of behavioral economics offers a promising and highly scalable approach to decreasing use of low-value services: asking clinicians to commit to avoid ordering such services and providing them and their patients with resources to support adherence to this commitment. This project will evaluate the effects of such an intervention across 2 large health systems, Michigan Medicine and IHA, through a mixed-methods, stepped wedge cluster randomized trial. In each of the study clinics, clinicians will be invited to commit to following a set of targeted Choosing Wisely® recommendations. Clinicians who make such a commitment, and their patients, will receive access to key resources to support adherence to this commitment. To measure the effects of the intervention, automated clinical data and medical record data before and after the intervention will be examined. Surveys and semi-structured interviews of both clinicians and patients will also be conducted to determine the effects of the intervention on their decision-making and experiences.

DETAILED DESCRIPTION:
A mixed-methods stepped wedge cluster randomized trial will be conducted in 8 primary care clinics of IHA, a private multispecialty group practice, and Michigan Medicine, a large academic health system. The study will test whether pre-encounter clinician commitments combined with patient and provider supports decrease overtreatment of type 2 diabetes among patients 65 and older, use of benzodiazepines and sedative-hypnotics among patients age 65 and older who have insomnia or anxiety, and use of PSA tests to screen for prostate cancer among men 75 and older. These 3 recommendations were chosen because they are commonly performed in primary care practice, have Choosing Wisely® recommendations against these low-value services, and represent situations in which clinician decisions about ordering of services can be unduly swayed by interactions with patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinician participants will be drawn from the pool of physicians, nurse practitioners, and physician assistants staffing the 8 primary care clinics.
* Patients of all 8 study clinics must meet criteria for one of the three Choosing Wisely® recommendations to be eligible to participate:

  * 65 and older with type 2 diabetes
  * 65 and older with insomnia and/or anxiety
  * male, 75 and older with no history of prostate cancer.

Exclusion Criteria:

* Patients who have cognitive impairment and/or a serious psychiatric diagnosis will not be eligible to participate in the surveys or interviews.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 489 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Difference in the proportion of intervention and control period visits with an applicable low-value treatment or test as specified by each respective Choosing Wisely® recommendation | 10 months
  The applicable low-value treatments or tests specified by the respective Choosing Wisely® recommendations are use of hypoglycemic medications for patients 65 years or older with diabetes and tight glycemic control, PSA testing among men 75 years or older with no history of prostate cancer, and use of benzodiazepine or sedative-hypnotic medications for patients with insomnia or anxiety who are 65 years or older.

SECONDARY OUTCOMES:
Patient trust in primary care provider | Within 1 week of primary care visit
  Self reported level of trust patient has in his or her primary care provider as measured by a 5-item scale.
Patient rating of provider | Within 1 week of primary care visit
  Patient's self-reported rating of their primary care provider as measured on a 0 to 10 scale.
Frequency of patient-provider conversations about the applicable low-value treatments or tests | Within 1 week of primary care visit
  Self-reported frequency of patient-provider conversations about the applicable low-value treatments or tests. The applicable low-value treatments or tests specified by the respective Choosing Wisely® recommendations are use of hypoglycemic medications for patients 65 years or older with diabetes and tight glycemic control, PSA testing among men 75 years or older with no history of prostate cancer, and use of benzodiazepine or sedative-hypnotic medications for patients with insomnia or anxiety who are 65 years or older.
Composite difference in the proportion of intervention and control period visits with an applicable low-value treatment or test as specified by each respective Choosing Wisely® recommendation | 10 months
  The study will combine data from all target recommendations (e.g., a composite outcome) where if one visit meets inclusion criteria for more than one target recommendation, they will be treated as independent visits.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey T. Kullgren, MS, MD, MPH, Principal Investigator — University of Michigan; Eve Kerr, MD, MPH, Principal Investigator — University of Michigan
Locations (9):
- United States (9):
  - IHA Family & Internal Medicine - West Arbor, Ann Arbor, Michigan
  - IHA Internal Medicine - Domino's Farms, Ann Arbor, Michigan
  - Michigan Medicine Briarwood Medical Group, Ann Arbor, Michigan
  - Michigan Medicine East Ann Arbor Health and Geriatrics Center, Ann Arbor, Michigan
  - University of Michigan Medical School, Ann Arbor, Michigan
  - Michigan Medicine Brighton Health Center, Brighton, Michigan
  - IHA Family & Internal Medicine - Cherry Hill, Canton, Michigan
  - Michigan Medicine Canton Health Center, Canton, Michigan
  - IHA Internal Medicine - Towsley, Ypsilanti, Michigan

REFERENCES:
- [Derived] Kullgren JT, Kim HM, Slowey M, Colbert J, Soyster B, Winston SA, Ryan K, Forman JH, Riba M, Krupka E, Kerr EA. Using Behavioral Economics to Reduce Low-Value Care Among Older Adults: A Cluster Randomized Clinical Trial. JAMA Intern Med. 2024 Mar 1;184(3):281-290. doi: 10.1001/jamainternmed.2023.7703. PMID 38285565